CLINICAL TRIAL: NCT02663466
Title: Importance of Erroneous Off-midline Closure as a Recurrence Factor in Limberg Flap Reconstruction in Sacrococcygeal Pilonidal Sinus: a Multicenter, Matched-case-control Study
Brief Title: Off-midline Closure Errors as a Risk Factor for Recurrence Following Limberg Flap in Patients With Pilonidal Sinus
Status: Completed | Type: Observational
Sponsor: Medical Park Gaziantep Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Kaplan, General Surgery, Medical Park Gaziantep Hospital
Other Study IDs: MK-005-PS
Record Dates: First submitted 2016-01-18; First posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Pilonidal Sinus; Recurrence
Keywords: pilonidal sinus; Limberg flap; off-midline closure concept; recurrence
MeSH Terms: conditions — Pilonidal Sinus; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Recurrent Group: Patients with clinically confirmed recurrence of sacrococcygeal pilonidal sinus following Limberg flap surgery were eligible (recurrent group, RG). They were evaluated for erroneous off-midline closures as an exposure variable.
  Interventions: Procedure: erroneous off-midline closures
- Nonrecurrent Group: Patients who underwent same surgery from the January 2008 to July 2015 but have not had recurrence in the five-year follow-up period (non-recurrent group, NRG) were accepted eligible. They were evaluated for erroneous off-midline closures as an exposure variable.
  Interventions: Procedure: erroneous off-midline closures

INTERVENTIONS:
Procedure: erroneous off-midline closures — All patients with pilonidal sinus recurrent disease following Limberg flap reconstruction in the recurrent group were examined by the authors in each study center and high resolution close-up photos of the patients' sacrococcygeal area were taken. These photos were then sent to all authors to asses and reach a collective decision to classify the erroneous off-midline closure technique and precisely measuring the distance between the flap border and the midline in the cleft. Same evaluation method was applied to the patients in nonrecurrent group. Following the completion of the assessments, all digital data of the patients were permanently deleted.
  Other Names: Rhomboid flap reconstruction

SUMMARY:
Background. Limberg flap, one of the recently being popularized off-midline closure techniques, is widely performed for the treatment of sacrococcygeal pilonidal sinus; however, recurrences still can be seen.

Objective. The aim of this study was to assess the relationship between recurrence and off-midline closure errors made in Limberg flap reconstructions.

Design. A multicenter, matched-case-control study was conducted in three participating centers in Turkey.

Settings. Each hospital's database was searched separately and all patients with and without recurrence who underwent LF surgery for primary SPS from January 2008 to July 2015 were identified.

Patients. Sixty patients with recurrent disease (recurrent group, RG) and 120 matched cases of recurrence-free patients for at least 5 years following surgery (non-recurrent group, NRG) were included to the study.

Interventions Main outcome measures. According to the off-midline closure concept, LF reconstructions were classified into incorrect closures (Type 1, 2 and 3) and correct closures (type 4, 5 and 6). Then the two groups were analyzed.

DETAILED DESCRIPTION:
Sacrococcygeal Pilonidal sinus (SPS) is a common disorder with estimated incidence of 1.1% in the community and 9% in soldiers. Pilonidal disease is a function of hair x force x vulnerability of the skin, the theory purposed by Karydakis in his article in 1992, and hair follicle obstruction and enlargement, assertion of Bascom are the most widely accepted explanation for etio-pathogenesis of the disease. It is such a disease that, there is still no clear consensus in regard to its gold-standard treatment modality, even though a lot of research and publications.

However, recently off-midline closure techniques has being popularized, by which the suture line is positioned off the midline to ensure minimal chance of recurrence. One of these techniques is the rhomboid, or Limberg, flap (LF) which is widely performed flap surgery for the treatment of SPS in Turkey. However, recurrences can be seen following wide excision and LF reconstruction; therefore, successful implementation of LF technique in the sacrococcygeal area requires well-known characteristics of the flap and problematic anatomy of the gluteal cleft.

There are many reports that favor Limberg flap over others. Although the authors also used to perform LF in patients with SPS with acceptable results until 2008, then they shifted their routine surgical preference to another off-midline closure technique for cosmetic reasons after this date. But increasingly more cases have administered to our institution due to the complications and recurrences after LF which performed elsewhere. Therefore the authors decided to investigate the technical reasons and risk factors of the problem to avoid complications and recurrence related to the incorrect flap design.

The authors first hypothesized that there are an association between erroneous off-midline closures and recurrence in patients underwent LF reconstruction for primary SPS. Then they designed a case-control study to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* age older than 16 years
* patients had been undergone LF reconstruction for primary SPS with no recurrence at least within the last 5 years
* patients with a clinical diagnosis of disease recurrence following LF surgery performed for primary SPS
* patients or his/her legal representative giving informed consent to make interview and participate to the study.

Exclusion Criteria:

* age younger than 16 years
* patients had been undergone a surgery other than LF for primary SPS
* patients with clinical history of multiple recurrence of the disease after any surgical procedure
* patients who had a recurrence due to the reasons other than correct or erroneous off-midline closure
* patients who had diabetes mellitus, or using steroids, had skin disorders such as hydradenitis suppurativa, had previously received phenol treatment, and patients who refused to give informed consent and who is unavailable or denied to make an interview.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with clinically confirmed recurrence of SPS following LF surgery (recurrent group, RG) and patients who underwent same surgery from the January 2008 to July 2015 but have not had recurrence in the five-year follow-up period (non-recurrent group, NRG) were accepted eligible.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
erroneous off-midline closures | within 1 mont after last patient included to the study
  Erroneous off-midline closure referred to the incision lines and/or angles of the LF are centered in- and/or crossed the midline or to be closer than 1 cm to the midline of the cleft between the buttocks.

SECONDARY OUTCOMES:
Suture type | within the first month after completion of the patient recruitment
  Suture type was referred to the LF skin suturing type. We classified suture types into two categories; i) intermittent type stitches with multifilament or monofilament sutures or with skin staplers, ii) continuous type which referred subcuticular stitch with a monofilament nonabsorbable suture.
Safe distance | within 1 month after the last patient included to the study
  Safe distance was referred the distance between the flap border and midline to be 1 cm or more.
Correct off-midline closures | within 1 month after last patient included to the study
  Proper off-midline closure referred to the incision lines and/or angles of the LF are not centered in- and/or not crossed the midline or to be farther than at least 1 centimeter to the midline of the cleft between the buttocks.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kaplan, M.D., Study Director — Bahcesehir University Medical School
Locations (1):
- Mehmet Kaplan, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No